CLINICAL TRIAL: NCT04182035
Title: Comparing the Effectiveness of Patient-tailored Treatment Versus Non Patient-tailored Treatment in Patients With Acute and Subacute Idiopathic Neck Pain
Brief Title: The Effectiveness of Patient-tailored Treatment in Patients With (Sub)Acute Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: B670201941044
Record Dates: First submitted 2019-11-12; First posted 2019-12-02 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Neck Pain; Acute Pain; Rehabilitation; Physical Therapy Modalities
Keywords: stratified care; patient-tailored therapy; subacute
MeSH Terms: conditions — Neck Pain; Acute Pain | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patient-tailored treatment group (Experimental): Objectives & approach: The subjects in the PTT group will receive the individual tailored treatment program combining best evidence active and passive treatment strategies (manual therapy, individual exercises) in combination with education tailored to the individual situation of the patient and selected home exercises. 9 individual therapy sessions will be performed, in combination with 9 additional home exercise sessions.. NRS and NDI-scores will be monitored before every treatment. The therapist will register when the cut-off score of 30% NDI reduction is present in order to determine the evolution in pain/disability reduction. The importance of self-efficacy will be emphasized and tailored home-exercises will be monitored and adjusted every week.
  Interventions: Other: patient-tailored therapy; Other: Education
- Non patient-tailored treatment group (Active Comparator): Objectives & approach: The NPTT will receive an individual (hands-off) treatment, which includes an active neck exercise program, non-tailored education and non-tailored home exercises, according to a previously published program with good results.53 The sessions will be performed once a week under supervision (9 therapy sessions, standard exercise program) and once a week by the patient at home (9 home exercise sessions, standard exercise program).
  Interventions: Other: Non-patient tailored therapy: generalized exercise program; Other: Education
- Control group (No Intervention): The subjects randomized to the control group will not receive any intervention, if necessary medication use is permitted and will be monitored using the iMTAQ. Patients will be asked not to seek other treatment options (if possible). If this is not possible, patients will be considered lost to follow-up.

INTERVENTIONS:
Other: patient-tailored therapy — The subjects in the PTT group will receive the individual tailored treatment program combining best evidence active and passive treatment strategies (manual therapy, individual exercises) in combination with education tailored to the individual situation of the patient and selected home exercises. 9 individual therapy sessions will be performed, in combination with 9 additional home exercise sessions.. NRS and NDI-scores will be monitored before every treatment. The therapist will register when the cut-off score of 30% NDI reduction is present in order to determine the evolution in pain/disability reduction. The importance of self-efficacy will be emphasized and tailored home-exercises will be monitored and adjusted every week.
  Arms: Patient-tailored treatment group
Other: Non-patient tailored therapy: generalized exercise program — The NPTT will receive an individual (hands-off) treatment, which includes an active neck exercise program, non-tailored education and non-tailored home exercises, according to a previously published program with good results.53 The sessions will be performed once a week under supervision (9 therapy sessions, standard exercise program) and once a week by the patient at home (9 home exercise sessions, standard exercise program).
  Arms: Non patient-tailored treatment group
Other: Education — Education considering neck pain information
  Arms: Non patient-tailored treatment group; Patient-tailored treatment group

SUMMARY:
The purpose of the present study is to examine if a patient-tailored treatment program has a better effect on pain and disability than a non-patient tailored treatment or wait and see approach in patients with (sub)acute (recurrent) NSNP. A secondary goal is to evaluate the global perceived effect, treatment adherence, recurrence, work absenteeism and medication use. All interventional treatment arms will consist of a treatment part in a clinical practice setting, under supervision of a trained physiotherapist, and an educational intervention and will be compared to the control group.

DETAILED DESCRIPTION:
Non-specific neck pain (NSNP) is a widespread health problems and a major cause of pain and disability. This condition is complex, disabling and has a heterogeneous presentation, which makes NSNP difficult to treat. Currently, the best evidence supports combining different forms of manual therapy (mobilizations, manipulations and manual muscle techniques), and exercises. Yet, identifying the most effective treatment characteristics and dosages remain challenging. Central in the debate about best practice management of NSNP and NSLBP is the efficacy of tailored versus generic (non-tailored) treatment. To date, sufficient evidence for the application of specific physiotherapy modalities or therapy aiming at specific NSNP subgroups is lacking. Although more research has already been conducted for the lumbar spine, there is an ongoing quest to identify relevant subgroups and provide patients with an assessment-driven targeted intervention to achieve meaningful and long-lasting changes.

Attempts have been made to identify relevant and homogeneous subgroups for patients with NSNP. Several classification systems have been proposed, based on (1) prognosis or (2) the underlying mechanism(s) driving the disorder: (2a) pain mechanisms, (2b) features of movement/posture/muscle activation , and (2c) pathology/diagnosis. The main goal of subgrouping patients is to enhance treatment efficiency. Nevertheless, a profound clinical reasoning process is necessary to identify clinically relevant subgroups. By identifying accurate and useful diagnostic criteria for NSNP and NSLBP, more informed decisions regarding the management of these conditions could be made.

Clinicians and researchers are hopeful that tailoring treatment to subgroups of patients may positively impact on patient outcomes and more efficient usage of health-care resources. For the lumbar spine, tailoring treatment to different subgroups is already present in literature. For example, in patients with pain provoked by postures/movements, tailoring treatment to modify specific features of posture/movement is effective and patients allocated to subgroups respond better to matched rather than unmatched interventions. Yet, other studies showed no additional benefit. Despite the growing interest for tailoring treatment for NSNP, the definition of tailored/stratified care is broadly used and interpretation is diverse. In order to determine best practice for the individual patient, tailoring the treatment should account for the multidimensional nature of non-specific spinal complaints and respect the individual characteristics of the patient within its subgroup. Additionally, it must take into account that patients may present with features of multiple subgroups or evolve through subgroups during treatments.

Previous studies on NSLBP already showed that targeting treatment can reduce costs and may improve outcomes when specific groups are compared. Unfortunately, at this moment, no conclusive high-quality evidence is present for its superiority. In addition to the lumbar spine, research on stratified care for NSNP is scarce compared to NSLBP research. Despite its major prevalence and socioeconomic consequences, no recommended or validated classification systems to stratify care for NSNP and to target specific subgroups are available. This suggests that the treatment decision in this heterogeneous group mostly depends on the clinical reasoning process, which is often incomplete in research on NSNP.

In order to evaluate the best practice for NSNP, a classification system based on a profound clinical reasoning process, identifying clinically relevant subgroups should be implemented to guide treatment tailoring and to allow a holistic and individual approach, instead of oversimplifying non-specific spinal complaints as one condition.

GOAL :

To evaluate the effectiveness of a patient tailored treatment (PTT) combined with individualized education, compared to (1) a non-patient tailored treatment (NPTT) consisting of a generalized exercise program with education and (2) a control group for (sub)acute (recurrent) nonspecific complaints.

ELIGIBILITY:
Inclusion Criteria:

* Non-specific neck pain, pain located in the cervico-thoracic and posterior shoulder region; without dominant arm pain.
* NDI scores score ≥10 % (more than no disability) and ≤68 % (less than complete disability)
* (Sub)acute complaints: <3 months
* Recurrent complaints but no neck pain episode the previous 3 months.
* Mean pain intensity scores: NRS > 3/10

Exclusion Criteria:

* Structural pathology, confirmed by imaging (disk herniation, nerve root compression, radiculopathy, severe rheumatoid diseases, fractures, traumatic alterations…) Shoulder pathology, vestibular pathology.
* Risk stratification: Startback tool for neck pain: high risk group
* BMI > 30 kg/m²
* Other cardiovascular/metabolic/systemic/ neurological diseases, fibromyalgia or chronic fatigue syndrome
* Psychiatric illnesses, history of depression, serious catastrophizing thoughts and/or low treatment expectations.[52]
* Chronic complaints (>3 months) or traumatic onset of the complaints
* Probable or definite neuropathic pain (according to the classification of Finnerup et al.)
* History of surgery in the head/neck or shoulder region
* Hypermobile patients
* Pregnancy or given birth in the preceding year.
* History of recurrent/chronic low back pain
* Primary headache

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Change in painscores in the neck region, overall pain score | Baseline, every supervised treatment (Week 1-9),follow up 3 weeks,3,6,12 months post treatment
  Numeric Rating Scale (score 0-10; 0=no pain; 10=worst pain)
Change in disability | Baseline, every supervised treatment (9x), follow up 3 weeks,3,6,12 months post treatment
  Neck Disability Index (score0-50; 0=no disability; 50=maximal disability)

SECONDARY OUTCOMES:
Change in Global Perceived Effect | After 3,6 & 9 supervised treatments, follow up 3 weeks,follow up 3,6,12 months
  Global Perceived Effect Scale (score:1-7; 1=a lot better, 7= a lot worse)
Change in medical costs | At baseline, follow up 3 weeks,3,6,12 months post treatment
  institute for Medical Technology Assessment (iMTA): Medical Costs Questionnaire
Change in productivity costs | At baseline, follow up 3 weeks,3,6,12 months post treatment
  institute for Medical Technology Assessment(iMTA): Productivity Costs Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Cagnie, Principal Investigator — UGent
Locations (1):
- Marjolein Chys, Ichtegem, België, Belgium

IPD SHARING:
Plan to Share IPD: No